CLINICAL TRIAL: NCT06887257
Title: RECOVER WITH INOCA: A Randomized, Prospective Study of a Cardiac Rehabilitation Program in Patients With Ischemia With Nonobstructive Coronary Artery Disease (INOCA)
Brief Title: RECOVER WITH INOCA: A Study of a Cardiac Rehabilitation Program in Patients With Ischemia With Nonobstructive Coronary Artery Disease (INOCA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: Spanish Society of Cardiology (Other)
Responsible Party: Principal Investigator, Margarita Calvo, Principal Investigator, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCB/2024/0926
Record Dates: First submitted 2025-03-14; First posted 2025-03-20 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: INOCA (Ischemia With Non Obstructive Coronary Artery Disease)
Keywords: INOCA; Cardiac rehabilitation; Functional capacity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cardiac rehabilitation group (treatment group) (Experimental): 3-mont telematic cardiac rehabilitation program for 3 months, including exercise, educational and psychological sessions
  Interventions: Other: Telematic cardiac rehabilitation program, that includes exercise, educational and psychological sessions during 3 months
- Standard recommendations (control group) (Active Comparator): Standard recommendations about exercise, education and psychological advise for INOCA patients
  Interventions: Other: Standard recommendations

INTERVENTIONS:
Other: Telematic cardiac rehabilitation program, that includes exercise, educational and psychological sessions during 3 months — 2 group and telematic exercise sessions/week, 1 educational session/week and 1 psychological session/week, during 3 months.
  There are no drugs or devices involved in the intervention.
  Arms: Cardiac rehabilitation group (treatment group)
Other: Standard recommendations — Standard recommendations about exercise, educational and psychologicla advice
  Arms: Standard recommendations (control group)

SUMMARY:
The goal of this clinical trial is to learn if a cardiac rehabilitation program (CRP) improves functional capacity in adults with INOCA (ischemia with non obstructive coronary arteries). The main questions it aims to answer are:

* Does CRP improves maximal functional capacity (measured by VO2peak) in INOCA patients?
* Does CRP improve as well quality of life, adherence to Mediterranean diet, emotional state, functional independence angina episodes and sleep quality?

Researchers will compare CRP (treatment group) to standard recommendations (control group) to see if CRP works better for INOCA patients

Participants will:

Take part of CRP or standard recommendations for 3 months Visit the clinic in the beginning and in the end of the study for checkups and tests

DETAILED DESCRIPTION:
A prospective, single-centre, randomized study with patients diagnosed with INOCA to assess their participation in a 3-month telehealth-based holistic cardiac rehabilitation program (CRP). Exclusion criteria were based on contraindications for participating in the telehealth CRP: alarm signs in the stress test (ventricular arrhythmias, hypotensive response, ST segment changes, or symptoms of ischemia), left ventricular ejection fraction (LVEF) <40%, or presence of pacemakers/defibrillators. Additionally, patients without a mobile device/tablet/computer with internet access to connect to exercise and educational sessions were excluded. Finally, participants should be stable in terms of angina episodes, defined as the absence of hospitalizations or decompensations in the number of angina episodes, as well as no changes in antianginal medications for 3 months prior to inclusion.

The primary endpoint is the improvement in functional capacity, objectively measured by the change in peak oxygen consumption (VO2peak) obtained from cardiopulmonary exercise testing (CPET) after 3 months of CRP (treatment group), compared to standard recommendations (control group). Secondary endpoints are CRP impact on quality of life, adherence to Mediterranean diet, emotional state, functional independence, angina episodes and sleep quality. The investigators selected pure VSA and pure MCA endotypes for the inclusion, to avoid confusion factors and to see if there were different results between both endotypes. A sample of 24 patients was selected to detect a 4.5 ml/kg/min difference in VO2peak.

The study scheme is as follows:

1. Recruitment: INOCA patients (confirmed diagnosis with microcirculation and provocation testing) are referred from ischemic heart disease consultations.
2. Initial Assessment Visit:

   * Part 1: Cardiologist and hemodynamic nurse explain the project, and if the patient agrees to participate, randomization (CRP yes or no) occur, and informed consent is signed. Blood samples are taken for initial assessment (basic profile, haemostasis, lipid profile, and HbA1c). Additionally, scales for quality of life (EuroQol), anxiety and depression (HADS), Mediterranean diet (PREDIMED), weekly exercise volume (IPAQ), functional (Barthel), and angina (SAQ-7) assessments are completed.
   * Part 2: Assessment in the cardiac rehabilitation clinic and initial CPET (cardiopulmonary stress test) testing for all patients. If the patient belongs to the CRP group, an individualized exercise prescription is made for the physiotherapist. If not, general exercise recommendations are provided. In both cases, a final CPET visit is scheduled at 3 months.
3. Cardiac Rehabilitation Program (3-month duration, for the intervention group): 2 individualized exercise sessions per week (via Teams platform) with the physiotherapist, 1 educational session per week via Teams with nursing, and 1 educational session per week via Teams with psychology.
4. Final Visit in Cardiac Rehabilitation: Scales wee reassessed, CPET is conducted, and a final medical assessment is performed. A final blood test and nursing assessment is also conducted, including an ad hoc patient experience survey regarding the program. A final medical report with their evolution and recommendations for follow up is given to all patients.

ELIGIBILITY:
Inclusion Criteria:

* All men or women >18 years old with cath lab diagnosis of INOCA of 2 possible endotypes: vasoespasm or microvascular disease.
* All participants must have a mobile device/tablet/computer with internet access to connect to exercise and educational sessions
* Participants should be stable in terms of angina episodes, defined as the absence of hospitalizations or decompensations in the number of angina episodes, as well as no changes in antianginal medications for 3 months prior to inclusion.

Exclusion Criteria:

* Alarm signs in the stress test (ventricular arrhythmias, hypotensive response, ST segment changes, or symptoms of ischemia)
* Left ventricular ejection fraction (LVEF) <40%, or presence of pacemakers/defibrillators

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
Maximal functional capacity | 3 months
  Change in VO2peak measured with CPET (cardiopulmonary stress test)

SECONDARY OUTCOMES:
EuroQol (EQ-5D) | 3 months
  * Full name: EuroQol Five-Dimension Scale
  * Purpose: Measures health-related quality of life (HRQoL) across five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. It also includes a visual analogue scale (VAS) for self-rated health.
  * Minimum value: 0 (equivalent to death) or negative values (worse than death, depending on country-specific value sets)
  * Maximum value: 1 (perfect health)
  * Interpretation: Higher scores indicate a better health-related quality of life.
PREDIMED | 3 months
  * Full name: PREDIMED Mediterranean Diet Adherence Screener
  * Purpose: Assesses adherence to the Mediterranean diet, which is associated with reduced cardiovascular risk and improved health outcomes.
  * Minimum value: 0 (no adherence)
  * Maximum value: 14 (maximum adherence)
  * Interpretation: Higher scores indicate a better outcome, meaning greater adherence to the Mediterranean diet and its associated health benefits. A score ≥9 suggests high adherence.
HADS | 3 months
  * Full name: Hospital Anxiety and Depression Scale - Depression (HADS-D) and Anxiety (HADS-A) Subscales
  * Purpose: Assesses symptoms of anxiety (HADS-A) and depression (HADS-D) in hospital and primary care settings, avoiding somatic symptoms to focus on emotional distress.
  * Minimum value: 0 (no symptoms)
  * Maximum value: 21 per subscale (total 42 if both are combined)
  * Interpretation: Higher scores indicate a worse outcome, meaning more severe anxiety or depression symptoms. Scores of 8-10 suggest mild symptoms, 11-14 moderate, and ≥15 severe symptoms.
Barthel Score | 3 months
  * Full name: Barthel Index of Activities of Daily Living
  * Purpose: Evaluates functional independence in activities of daily living (ADLs), such as bathing, dressing, mobility, and feeding, primarily in stroke and rehabilitation patients.
  * Minimum value: 0 (total dependence)
  * Maximum value: 100 (complete independence)
  * Interpretation: Higher scores indicate a better outcome, meaning greater independence in daily activities.
Angina episodes | 3 months
  Change in the number of angina episodes/month
PSQI | 3 months
  * Full name: Pittsburgh Sleep Quality Index
  * Purpose: Assesses sleep quality and disturbances over a 1-month period. It consists of 7 components: Subjective sleep quality, Sleep latency, Sleep duration, Habitual sleep efficiency, Sleep disturbances, Use of sleep medication, Daytime dysfunction
  * Minimum value: 0 (best sleep quality)
  * Maximum value: 21 (worst sleep quality)
  * Interpretation: Higher scores indicate a worse outcome, meaning poorer sleep quality. A global PSQI score >5 suggests poor sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Margarita Calvo-Lopez, MD, Principal Investigator — Hospital Clinic of Barcelona
Locations (1):
- Villarroel 170, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
All IPD collected throughout the trial
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Beginning 3 months and ending 1 year after the publication of results
Access Criteria: Access to IPD and supporting information will be granted to qualified researchers, healthcare professionals, and regulatory authorities for scientific, clinical, or public health purposes. Requests will be reviewed by an independent data access committee to ensure compliance with ethical and legal requirements.
  Available Data: De-identified IPD, study protocol, statistical analysis plan, informed consent form template, and study results summary.
  Access Mechanism: Applicants must submit a research proposal, sign a data use agreement (DUA), obtain committee approval, and access data via a secure platform.
  Ethical and Legal Compliance: Access will follow GDPR, HIPAA, and ethical guidelines, ensuring de-identification and restricted use for approved research purposes.
  Data Availability: Data will be accessible for at least five years post-publication, with potential extensions.
  Contact: For access requests, contact margacal1912@gmail.com